CLINICAL TRIAL: NCT04007627
Title: Dose Reduction and Acquisition Parameters Optimization for PEDiatric Digital Radiography
Acronym: DRAPOPED
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 19CAM-DRAPOPED
Record Dates: First submitted 2019-06-18; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Pediatric Radiology
Keywords: ALADA; IQ; Pediatric Radiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To reduce "As Low As Diagnostically Acceptable" (ALADA) the X ray exposure of pediatric radiology by using a new post treatment processing algorithm (S-Vue, Samsung table GC85A).

DETAILED DESCRIPTION:
The study will investigate the minimum dose required to obtain acceptable image quality for different pediatric localizations (abdomen, thorax, pelvis, spine) by using a simulation tool of different dose levels. Three different radiologists blinded to the simulated dose level will score the images independently by using a dedicated image quality scoring grid.

ELIGIBILITY:
Inclusion Criteria:

* Children aged under 18 years and under 80 kg;
* Prior radiography perfomed within 6 months before the beginning of the study.

Exclusion Criteria:

- Refusal of parents to participate to the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric population
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Assesment of image quality by radiologists blinded to the simulated dose level | through study completion, an average of 6 months
  Three different radiologists will score the images of localizations of abdomen, thorax, pelvis, spine independently by using a dedicated image quality scoring grid.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Adamsbaum, MD, PhD, Principal Investigator — Faculté de Médecine Paris Sud, Service de Radiologie Pédiatrique, C.H.U. Bicêtre; Joëlle Feghali, MS, Study Director — Service de Radiologie Pédiatrique, C.H.U. Bicêtre
Locations (1):
- Service de Radiologie Pédiatrique, C.H.U. Bicêtre, APHP, Le Kremlin-Bicêtre, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No